CLINICAL TRIAL: NCT05331872
Title: A Phase I, Open-label Trial on the Safety and Efficacy of Human Umbilical Cord-derived Mesenchymal Stem Cell Administration in the Management of Adult Liver Cirrhosis
Brief Title: Umbilical Cord-derived Mesenchymal Stem Cell Infusion in the Management of Adult Liver Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC.19.29
Record Dates: First submitted 2022-04-06; First posted 2022-04-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human umbilical cord-derived mesenchymal stem cell transplantation for patients with liver cirrhosis (Experimental): Umbilical cords from healthy donor are processed with 24 hours after vaginal delivery.
  The cords are delivered in a sterilized jar the laboratory to process. After washing in PBS to remove any contaminating blood, the cord is cut into small pieces. The pieces are minced and digested by enzyme. The UC-MSCs is cultured and expanded using commercially available serum-free and xeno-free medium at 37°C in a humidified atmosphere with 5% CO2. The UC-MSCs is suspended in 15 ml of saline buffer
  Interventions: Biological: Human umbilical cord-derived mesenchymal stem cell infusion

INTERVENTIONS:
Biological: Human umbilical cord-derived mesenchymal stem cell infusion — Human umbilical cord-derived mesenchymal stem cell infusion in the management of adult liver cirrhosis

SUMMARY:
This is a phase I, open label, single arm trial using UC-MSCs to treat patients with liver cirrhosis that includes 20 patients. The primary outcome measure will be change in MELD score at 3, 6, and 12 months after UC-MSC transplantation from baseline. The safety is assessed by frequency and severity of the adverse event or serious adverse event associated with stem cell injection. This study could reconfirm the efficacy of stem cell transplantation for liver cirrhosis and would open a novel cell therapy for the treatment of adult liver cirrhosis.

DETAILED DESCRIPTION:
Liver cirrhosis is defined as the histological development of regenerative nodules surrounded by fibrous bands and causes by many forms of liver diseases and conditions such as hepatitis and chronic alcoholism. Liver cirrhosis has become one of the major causes of morbidity and mortality with over one million people died due to cirrhosis in 2010 worldwide. Currently, the only curative treatment for end-stage liver disease is liver transplantation. However, the shortage in donor organ availability and the side-effect associated with long-term immunosuppression after transplant requires the development of new alternative therapies for liver cirrhosis. Recent clinical trials demonstrate that bone marrow-derived stem cells (BMDSCs) as well as umbilical cord-derive mesenchymal stem cells (UC-MSCs) improve liver function in patients with liver cirrhosis. In Vietnam, however, there are no clinical trials to date that investigate the potential of UC-MSCs for liver cirrhosis management. This is a phase I, open label, single arm trial using UC-MSCs to treat patients with liver cirrhosis that includes 20 patients. The primary outcome measure will be change in MELD score at 3, 6, and 12 months after UC-MSC transplantation from baseline. The safety is assessed by frequency and severity of the adverse event or serious adverse event associated with stem cell injection. This study could reconfirm the efficacy of stem cell transplantation for liver cirrhosis and would open a novel cell therapy for the treatment of adult liver cirrhosis

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old.
* Patients diagnosed of liver cirrhosis: splenomegaly, elevated hepatic enzymes and/or esophageal varices detected by endoscopy, or liver biopsy demonstrated liver cirrhosis
* Be willing to complete the study and sign the consent form.

Exclusion Criteria:

* Younger than 18 or older than 70 years old
* Recent infection
* Patients with history of chronic diseases such as cancer, chronic hepatitis, chronic kidney disease.
* Any clinically significant blood coagulation disorder(s)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events and serious adverse events (AEs or SAEs) | up to the 12-month period following the first UC-MSCs infusion
  To assess safety: the number of AEs or SAEs during and after allogenic umbilical cord-mesenchymal stem cells (UC-MSCs) infusion

SECONDARY OUTCOMES:
Change of liver function through the Model for End Stage Liver Disease (MELD) score | 3 months, 6 months, 12 months after the UC-MSCs infusion
  The MELD score is negatively correlated with the liver function, in which higher scores indicative a poorer liver function. The MELD score decrease show clinical improvement. The MELD score is calculated using the following formula:
  MELD score = 10 * (0.957 ln (serum creatinine, mg/dl) + 0.378 ln (bilirubin, mg/dl) +1.12 ln (INR) + 0.643).
Change in health-related quality of life using Chronic Liver Disease Questionnaire - (CLDQ) | 3 months, 6 months, 12 months after the UC-MSCs infusion
  CLDQ was developed to evaluate the impact of chronic liver diseases (CLD) on quality of life. The CLDQ includes 29 items in the following domains: abdominal symptoms, fatigue, systemic symptoms, activity, emotional function and worry. The scores range from 1 to 7, whit higher values indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Liem Nguyen, PHD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No